CLINICAL TRIAL: NCT06059950
Title: Examining the Feasibility of the Mindfulness Flow Program (MFP) on Archers
Brief Title: Feasibility of the Mindfulness Flow Program (MFP) on Archers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Lo Ka Kay Cynthia, PhD student, Hong Kong Metropolitan University, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKMetU20210320
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Flow Program (Experimental): Mindfulness flow program, with 11 sessions conducted via Zoom video meeting and one in-person session of sport-specific session.
  Interventions: Behavioral: Mindfulness Flow Program

INTERVENTIONS:
Behavioral: Mindfulness Flow Program — The mindfulness flow program (MFP) consisted of eleven 60-minute sessions via Zoom, with one session per week. Additionally, a 120-minute in-person sport-specific session were conducted.

SUMMARY:
Mindfulness-based interventions have gained popularity among elite athletes, but their effectiveness for enhancing archery performance remains inconsistent. This study examined the feasibility of a 12-week mindfulness flow program (MFP) specifically designed for archers, and assessed the effect of the MFP on shooting performance. The intervention aims to enhance shooting performance, mindfulness, and the flow state, while reducing post-intervention anxiety.

DETAILED DESCRIPTION:
The primary goal of the present study was to test the feasibility of a prototype mindfulness flow program (MFP), with 11 sessions conducted via Zoom video meeting and one in-person session of sport-specific session. Additionally, the program seeks to examine the psychological outcomes associated with the intervention specifically among archery athletes. It is anticipated that the experimental group will show reduced anxiety levels and increased levels of mindfulness and flow when comparing their baseline and post-intervention assessments. This study explores the potential of delivering mindfulness programs conveniently to sport populations via the internet, supplemented by one face-to-face sport-specific session to enhance mindfulness and improve sports performance among athletes.

ELIGIBILITY:
Inclusion Criteria:

* at least one year of archery training experience and training for at least two hours per week

Exclusion Criteria:

* Participants who had previously participated in a mindfulness session were excluded

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-09-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Mindfulness Flow Program (MFP) | up to two weeks
  To assess the feasibility of the MFP, the athletes completed a feedback evaluation questionnaire adapted from Kuyken immediately after the end of the intervention (Kuyken et al., 2013). The questionnaire included questions about the number of sessions attended, the frequency of mindfulness practice after class, and the likelihood of continuing to use what they had learned from the course and of introducing the course to other athletes. The athletes rated their enjoyment of each session, on a 10-point Likert scale ranging from 1 (strongly disliked) to 10 (strongly liked).

SECONDARY OUTCOMES:
Shooting scores | up to 20 weeks
  Shooting scores was assessed using the World Archery Federation's qualifying competition procedures (World Archery Federation, 2022). All of the shooters were required to complete 72 shots. The total scores for the 72 shots were used for further analysis. Higher total scores indicated better shooting performance.
Cognitive State Anxiety | up to 20 weeks
  Cognitive state anxiety was assessed using the the Chinese Version (Cox et al., 2003) of the Competitive State Anxiety Inventory-2 Questionnaire (CSAI-2; Martens et al., 1990). The cognitive state anxiety scale consisted of nine items. Each item was scored on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much so). Higher scores indicate higher cognitive state anxiety level.
Somatic State Anxiety | up to 20 weeks
  Somatic state anxiety was assessed using the Chinese Version (Cox et al., 2003) of the Competitive State Anxiety Inventory-2 Questionnaire (CSAI-2; Martens et al., 1990). The somatic state anxiety scale consisted of nine items. Each item was scored on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much so). Higher scores indicate higher somatic state anxiety level.
Self-confidence | up to 20 weeks
  Self-confidence was assessed using the Chinese Version (Cox et al., 2003) of the Competitive State Anxiety Inventory-2 Questionnaire (CSAI-2; Martens et al., 1990). The self-confidence scale consisted of nine items. Each item was scored on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much so). Higher scores indicate higher self-confidence level.
Mindfulness | up to 20 weeks
  Mindfulness were assessed using the Chinese version (Deng et al., 2011) of Five facets mindfulness questionnaire (FFMQ) (Baer et al., 2006), with 39 items scored on a 5-point Likert scale (1 = never or very rarely true; 5 = very often or always true). Higher scores indicate higher mindfulness level
Flow state | up to 20 weeks
  Flow state was assessed using the Chinese Version (Liu, 2010) of the Short Dispositional Flow Scale (SDFS; Jackson et al., 2008). The nine SDFS items were scored on a 5-point Likert scale ranging from 1 (never) to 5 (always), where a higher score indicates a higher overall flow state.

CONTACTS AND LOCATIONS:
Overall Officials: Mum Yee Tse, PhD, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Lion Rock Archery Venue, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No